CLINICAL TRIAL: NCT00851461
Title: Effect of Goserelin (Zoladex®) in Spinal and Bulbar Muscular Atrophy in Thai Patients
Brief Title: Effect of Goserelin (Zoladex®) in Spinal and Bulbar Muscular Atrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Dean of Ramathibodi Hospital, Faculty of Medicine, Ramathibodi Hospital, Bangkok, Thailand
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID11-50-17
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2009-02

CONDITIONS: Spinobulbar Muscular Atrophy; Kennedy's Disease
Keywords: Spinobulbar muscular atrophy; Kennedy's disease; Goserelin; Electrophysiologic study; Inclusion body
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Goserelin — Goserelin 10.8 mg SC every 3 months
  Other Names: Zoladex LA
Procedure: Electrophysiologic study — Nerve conduction study Electromyogram
  Other Names: NCV; EMG
Procedure: tissue biopsy — skin and muscle biopsy before and after treatment every year

SUMMARY:
This is a therapeutic trial study to demonstrate whether Goserelin, a LHRH agonist has benefit in SBMA

Objective:

1. To study effects of Goserelin to clinical course of patients with spinal and bulbar muscular atrophy in Thailand
2. To demonstrate physiological and pathological changes in treated patients with Goserelin.
3. To assess tolerability and adverse effect of Goserelin therapy

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Males, age over 20 years, undesired fertility
3. Have positive family history of muscle weakness with these clinical signs:

   * bulbar involvement (difficulty in breathing, swallowing, talking)
   * muscle atrophy with or without fasciculation
   * decrease or normal deep tendon reflex
   * normal Babinski response
   * no sensory impairment
   * mild tremor (either postural or intention)
   * gynecomastia
   * decrease libido and infertility
4. Subjects have a confirmed diagnosis to SBMA by both NCV test and DNA study demonstrated the number of CAG repeated more than 35.

Exclusion Criteria:

1. Have weakness caused by other etiologies and have liver or kidney disease.
2. Have currently prostatic cancer
3. Want to have a child
4. Participation in a clinical study during the last 30 days.
5. Females and children age < 20 years old

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2011-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
muscle power | every 3 months

SECONDARY OUTCOMES:
electrophysiologic study (Nerve conduction and Electromyogram) | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Thanyachau Sura, M.D., MRCP, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Medical Genetics and Molecular Medicine Unit,, Department of Medicine, Ramathibodi Hospital, Bangkok, Bangkok, Thailand